CLINICAL TRIAL: NCT01347671
Title: A Randomized 4-week Phase IIa Trial Evaluating the Efficacy, Safety, and Tolerability of GRT6005, a New Centrally Acting Analgesic, in Subjects With Pain Due to Diabetic Polyneuropathy.
Brief Title: Safety and Efficacy of GRT6005 in Pain Due to Diabetic Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 430409; 2010-022557-42 (EudraCT Number)
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pain; Diabetic Neuropathies
Keywords: analgesia; analgesics; pain; chronic pain; neuropathic pain
MeSH Terms: conditions — Pain; Diabetic Neuropathies; Agnosia; Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 25 µg GRT6005 (Active Comparator): Participants allocated to this treatment arm will receive a daily dose of 25 µg GRT6005 per day
  Interventions: Drug: GRT6005
- 75 µg GRT6005 (Active Comparator): Participants allocated to this treatment arm will receive a daily dose of 75 µg GRT6005 per day
  Interventions: Drug: GRT6005
- 200 µg GRT6005 (Active Comparator): Participants allocated to this treatment arm will receive a daily dose of 200 µg GRT6005 per day
  Interventions: Drug: GRT6005
- Matching Placebo (Placebo Comparator): Participants allocated to this treatment arm will receive a dose of matched placebo once a day.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: GRT6005 — 25µg/day once daily
  Arms: 25 µg GRT6005
Drug: GRT6005 — 75 µg/day once daily
  Arms: 75 µg GRT6005
Drug: GRT6005 — 200 µg/day once daily
  Arms: 200 µg GRT6005
Drug: Matching Placebo — Once daily
  Arms: Matching Placebo

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of GRT6005 in patients with painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 to 75 years old.
* Type 1 or type 2 diabetes.
* Painful DPN symptoms and signs for at least 3 months.
* Blood glucose controlled with medication.
* Glycosylated hemoglobin not greater than 9.5 or 11%, country dependent.
* Prior analgesic medication.
* Average score of 4 or greater on the 11 point NRS during the last 3 days prior to randomization.

Exclusion Criteria:

* Impaired liver, cardiac or renal function.
* Breastfeeding and pregnancy.
* History of substance abuse, alcohol or medication.
* Chronic gastrointestinal disease.
* History of seizures and or epilepsy.
* History or presence of malignancy.
* Presence of painful medical conditions that are not due to diabetic neuropathy, e.g. rheumatoid arthritis.
* Allergies to opioids, acetaminophen or excipients of the medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in mean daily pain intensity score | Baseline to Week 4
  Participants will be selected based on their medical history and clinical examination.
  Efficacy of the treatment (i.e., reduction of pain) will be evaluated with the 11-point numeric rating scale (NRS), where 0 represents no pain and 10 represents "pain as bad as you can imagine".

SECONDARY OUTCOMES:
Response measured in percentage change of pain intensity from baseline | End of 4 Weeks
Changes in Quantitative Sensory Testing from baseline | Baseline, week 1 and week 4
Neuropathic Pain Scale, changes from baseline | End of 4 weeks
Short Form of the Brief Pain Inventory, changes from baseline | End of 4 weeks
Leeds Sleep Evaluation Questionnaire | End of treatment
Quality of Life Index -Short-Form-12®, from baseline | End of treatment
Patient's Global Impression of Change | End of treatment
Quality of Life EuroQoL-5 Dimension score, change from baseline | End of 4 weeks
Rescue medication use | End of 4 weeks
Clinical Opioid Withdrawal Scale | End of 4 weeks
Plasma concentration | End of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, Prof. Dr., Principal Investigator — ikfe GmbH, Institut for Klinische Forschung und Entwicklung, Parcusstr. 8, 55116 Mainz, Germany
Locations (22):
- Site 4502, Sofia, Bulgaria
- Germany (16):
  - Site 4112, Aschaffenburg
  - Site 4109, Bad Oeynhausen
  - Site 4101, Berlin
  - Site 4110, Berlin
  - Site 4111, Dresden
  - Site 4107, Hamburg
  - Site 4117, Hamburg
  - Site 4108, Hanover
  - Site 4104, Hanover
  - Site 4115, Heidelberg
  - Site 4106, Kiel
  - Site 4102, Lübeck
  - Site 4103, Mainz
  - Site 4105, Münster
  - Site 4113, Schwerin
  - Site 4116, Wangen
- Romania (5):
  - Site 4405, Bucharest
  - Site 4402, Bucharest
  - Site 4407, Sibiu
  - Site 4401, Târgu Mureş
  - Site 4406, Timișoara